CLINICAL TRIAL: NCT06895278
Title: Evaluation of Articular Damage in Patients With Juvenile Idiopathic Arthritis (JIA) After Transition to Adult Care and Correlation With Disease Characteristics and Treatments.
Brief Title: Articular Damage in Patients With Juvenile Idiopathic Arthritis After Transition to Adult Care
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 35/24; 1709 (Registry Identifier: Registro degli Studi Osservazionali (RSO))
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Juvenile Chronic Arthritis
Keywords: Juvenile idiopathic arthritis; JIA; transition to adult; articular damage
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Methotrexate; Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Methotrexate group: Patients who underwent transition from pediatric to adult rheumatology care who spent most of their disease time on methotrexate therapy
  Interventions: Drug: Methotrexate
- Biologic therapy group: Patients who underwent transition from pediatric to adult rheumatology care who spent most of their disease time on biologic therapy
  Interventions: Drug: Biological Drug

INTERVENTIONS:
Drug: Methotrexate — Prevalent use of methotrexate in pediatric age
  Groups: Methotrexate group
Drug: Biological Drug — Prevalent use of biological drugs in pediatric age
  Groups: Biologic therapy group

SUMMARY:
Juvenile idiopathic arthritis (JIA) is the most common childhood chronic rheumatic disease, encompassing all forms of arthritis that persist for more than 6 weeks, with onset before age 16, after exclusion of other causes of arthritis. It is a heterogeneous disease, whose complexity is only partially encompassed by the actual classification criteria and it is characterized by prolonged synovial inflammation that can lead to joint destruction.

Whilst the assessment of structural joint damage is part of the routinary evaluation of disease severity and progression in patients with rheumatoid arthritis (RA), to the extent that it is considered a key end-point outcome in treatment efficacy studies, this is not the same for JIA. Some recommendations have been elaborated based on expert opinion, but only recently they have been translated into clinical practice. Such a discrepancy in approaching chronic arthritis has been for many years due to the lack of articular damage radiographic scoring system validated for pediatric age. Actually, joint space narrowing, bone erosions and demineralization, which is typical of adult articular damage, are not the same changes observed in pediatric population where early growth plate closure, epiphyseal deformity and growth asymmetries can be the major signs.

The transition process from the pediatric to the adult health care team is a critical moment in the clinical history of patients with JIA, often hampered by the absence of specific criteria for the assessment of disease activity, the lack of specific treatment recommendations for JIA adult patients, the poor adolescent-specific training for adult rheumatologists, and the lack of communication between pediatric and adult centers. Adult patients with JIA have their own specific identity and should not be inappropriately re-categorized as having RA, ankylosing spondylitis or another condition once transitioned to the adult rheumatologist.

The aim of this study is to quantify the articular damage of adult patient with JIA after closure of growth plates. This represent a sort of starting burden carried by the patients who receive transition to the adult rheumatologist care and which should be minimized in order to reduce long-term complications. Furthermore, the study aims to analyze possible correlations between the presence of articular damage, therapies taken in pediatric age, and characteristics of JIA at the onset and during the clinical course of the disease

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 16 to 25 years who received a diagnosis of JIA in pediatric age according to International League of Associations for Rheumatology criteria (2001) and who have begun the process of transition to adult care.
2. Young adults undergoing healthcare transition process from the the pediatric to adult rheumatology since 2016.
3. Patients with radiological evidence of joint plates closure.
4. X-ray images of hands, hips, and knees available

Exclusion Criteria:

1. Patients cared at the adult rheumatology clinic who received a diagnosis of arthritis in the adult age.
2. Patients with other orthopedic conditions or affected by other diseases leading to osteoporosis or skeletal deformities.
3. Patients affected by other rheumatological conditions who underwent healthcare transition process from the the pediatric to adult rheumatology center.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients with Juvenile Idiopathic Arthritis who started transition process from a pediatric to an adult rheumatology center in the last 10 years will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean difference between groups in the radiographic Sharp/Van der Heijde score | At transition from pediatric to adult care, on average at the age of 18
  Radiological examinations of small joints (hands/wrists) will be pseudo-anonymized and centralized to a blinded radiologist to evaluate damage using the Sharp/Van der Heijde score, evaluating joint space narrowing and erosion with a range from 0 to 4 and from 0 to 5, respectively. The total Sharp/van der Heijde score is calculated as the sum of the scores for joint space narrowing (range 0-120) and erosion (range 0-160) and ranges from 0 to 280.
Mean difference between groups in the radiographic Larsen score | At transition from pediatric to adult care, on average at the age of 18
  Radiological examinations of knees and hips will be pseudo-anonymized and centralized to a blinded radiologist to evaluate damage using the Larsen score. The grading scale ranges from 0 to 5 (0=intact bony outlines and normal joint space, 5=mutilating changes). The Larsen score ranges from 0 to 120.

SECONDARY OUTCOMES:
Associations between the radiographic Sharp/Van der Heijde score and clinical characteristics | At transition from pediatric to adult care, on average at the age of 18
  The following variables will be included in multivariate analysis: age, age at onset, gender, family history of autoimmunity; clinical features of the disease during pediatric age (i.e., number and type of involved joints, JIA category according to 2001 International League of Associations for Rheumatology classification criteria, presence of enthesitis, tenosynovitis, psoriasis and uveitis in the patients' history); laboratory data (i.e., blood count, inflammation indexes, immunoglobulin levels, predisposing HLA, antinuclear antibodies, rheumatoid factor; disease activity score (JADAS-27 score) in the period closest to the radiography execution; therapies taken during the pediatric disease course.
Associations between the radiographic Larsen score and clinical characteristics | At transition from pediatric to adult care, on average at the age of 18
  The following variables will be included in multivariate analysis: age, age at onset, gender, family history of autoimmunity; clinical features of the disease during pediatric age (i.e., number and type of involved joints, JIA category according to 2001 International League of Associations for Rheumatology classification criteria, presence of enthesitis, tenosynovitis, psoriasis and uveitis in the patients' history); laboratory data (i.e., blood count, inflammation indexes, immunoglobulin levels, predisposing HLA, antinuclear antibodies, rheumatoid factor; disease activity score (JADAS-27 score) in the period closest to the radiography execution; therapies taken during the pediatric disease course.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Azienda sanitaria di Reggio Emilia - Arcispedale Santa Maria Nuova, Reggio Emilia, Italia
  - IRCCS Materno Infantile "Burlo Garofolo", Trieste, Italia
  - Istituto Azienda sanitaria universitaria Friuli Occidentale - Ospedale "Santa Maria della Misericordia", Udine, Italia

IPD SHARING:
Plan to Share IPD: No